CLINICAL TRIAL: NCT06455670
Title: Effects of Chinese Medicine on Patients With Severe Acute Exacerbation of COPD：A Multicentre, Randomised, Double-blind, Placebo-parallel Controlled Trial
Brief Title: Effects of Chinese Medicine on Patients With Severe Acute Exacerbation of COPD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henan University of Traditional Chinese Medicine (Other)
Collaborators: Peking University Third Hospital (Other); Jiangsu Province Hospital of Traditional Chinese Medicine (Other); Chengdu University of Traditional Chinese Medicine (Other); Affiliated Hospital of Liaoning University of Traditional Chinese Medicine (Other); Shenzhen Hospital of Southern Medical University (Other); Qingdao Haici Hospital (Other); Xiangyang Hospital of Traditional Chinese Medicine (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CM for Severe AECOPD
Record Dates: First submitted 2024-05-28; First posted 2024-06-12 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Acute Exacerbation Of Chronic Obstructive Pulmonary Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chinese medicine granules plus western medicine treatment (Experimental): On the basis of conventional western medicine treatment, the experimental group will be given Sanhan Huayin granule , Qingre Huatan granule or Zaoshi Huatan granule based on CM syndrome differentiation.Take 1 dose daily for 10 days.
  Interventions: Drug: Sanhan Huayin recipe, Qingre Huatan recipe or Zaoshi Huatan recipe
- Chinese medicine granules placebo plus western medicine treatment (Placebo Comparator): On the basis of conventional treatment of western medicine, in the experimental group 5% of the placebo drug, color, smell, taste, appearance, weight, similar to the experimental drug, drug packaging and test group. One dose was given daily for 10 days.
  Interventions: Drug: Sanhan Huayin recipe placebo, Qingre Huatan recipe placebo or Zaoshi Huatan recipe placebo

INTERVENTIONS:
Drug: Sanhan Huayin recipe, Qingre Huatan recipe or Zaoshi Huatan recipe — On the basis of conventional treatment of western medicine,the experimental group will be given Sanhan Huayin granule , Qingre Huatan granule or Zaoshi Huatan granule based on CM syndrome differentiation.Take 1 dose daily for 10 days.
  Arms: Chinese medicine granules plus western medicine treatment
Drug: Sanhan Huayin recipe placebo, Qingre Huatan recipe placebo or Zaoshi Huatan recipe placebo — On the basis of conventional treatment of western medicine, in the experimental group 5% of the placebo drug, color, smell, taste, appearance, weight, similar to the experimental drug, drug packaging and test group. One dose was given daily for 10 days.
  Arms: Chinese medicine granules placebo plus western medicine treatment

SUMMARY:
The purpose of this study was to evaluate the effects of Chinese Medicine on patients with severe AECOPD, and to provide a basis for the establishment of integrated CM and Western medicine diagnosis and treatment scheme for patients with severe AECOPD.

DETAILED DESCRIPTION:
Aiming at the key problems such as the lack of high-quality clinical research evidence of Chinese medicine in the prevention and treatment of severe AECOPD, this study adopted a multi-center, randomized, double-blind, placebo-controlled parallel trial design, taking 468 severe AECOPD patients as the research object, to evaluate the clinical efficacy and safety of Chinese medicine combined with western medicine in the treatment of severe AECOPD. To establish an integrated Chinese and western medicine diagnosis and treatment plan to reduce the treatment failure rate of severe AECOPD patients, and to form high-level evidence-based evidence.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with severe AECOPD.;
2. Age 40-80 years old;
3. Chinese medicine diagnosis consistent with external cold and internal drink syndrome, or phlegm-heat congestion of the lungs syndrome, or phlegm turbidity obstruction of the lungs syndrome;
4. Voluntarily accept the treatment and sign the informed consent form;

Exclusion Criteria:

1. Pregnant and lactating women.
2. delirious, dementia, various mental patients and other people who cannot communicate normally.
3. Patients with severe cardiac insufficiency (NYHA grade IV), malignant arrhythmia and hemodynamic instability.
4. Patients with acute respiratory failure who require tracheal intubation or invasive mechanical ventilation.
5. Complicated with bronchiectasis, active tuberculosis, severe liver and kidney disease (severe liver disease refers to cirrhosis, portal hypertension and varicose vein bleeding, etc., serious kidney disease including dialysis, kidney transplantation, etc.), pneumonia, HIV infection or immunosuppressive state, advanced malignant tumor, etc.
6. long-term bedridden patients for various reasons.
7. Out-of-hospital treatment for more than 3 days.
8. Participate in other drug clinical investigators within 1 month before enrollment.
9. Allergic to therapeutic drugs.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 468 (Estimated)
Dates: Start 2024-10-20 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Treatment failure rate | During the 10 days treatment period and the 3 months follow-up period.
  The number of treatment failures in both groups during the study period was measured. Treatment failure was defined as the following: (1) the need for or receipt of tracheal intubation or invasive mechanical ventilation during hospitalization, or (2) the need for or transfer to an intensive care unit during hospitalization, or (3) the duration of hospitalization for the current acute exacerbation of COPD for more than 14 days, or (4) death during hospitalization or within 30 days after discharge, or (5) readmission for an acute exacerbation of COPD within 30 days after discharge.

SECONDARY OUTCOMES:
The COPD Assessment Test(CAT) | Changes in baseline CAT scores at day 10 of the treatment period and at 1 and 3 months of follow-up.
  The COPD Assessment Test (CAT) is an 8-item questionnaire that assesses health status in patients with COPD. The questionnaire uses a 0-5 point scale, with higher values indicating a greater impact of COPD on the patient.
The number and severity of acute exacerbations | Within 3 months of follow-up period.
  The number and severity of acute exacerbations during the follow-up period.
Readmission rate of acute exacerbations | Within 3 months of follow-up period.
  The number of readmissions due to acute exacerbations during the follow-up period.
The time to the first exacerbation of COPD | Within 3 months of follow-up period.
  The time to the first COPD exacerbation during the study period.
Dyspnea score | Changes in baseline mMRC scores at days 4, 7, and 10 of the treatment period and at 1 and 3 months of follow-up.
  The modified Medical Research Council dyspnoea scale (mMRC) will be used to assess severity of dyspnea. The mMRC scale is a 4-point (0-4) scale. "0" means no dyspnea perception, "4" means severe dyspnea perception.
COPD Acute exacerbation tool (EXACT) score | 0 and 10 days in the treatment period, 1 and 3 months in the follow-up period.
  The EXAcerbations of Chronic Pulmonary Disease Tool (EXACT) is a questionnaire that assesses symptoms in patients with COPD. The questionnaire is on a scale from 0 to 5, with higher values indicating a greater impact of COPD on the patient.
Length of hospital stay | During the 10 days treatment period and the 3 months follow-up period.
  Through study /treatment phase completion,an average of 10 days.
Antibacterial application time | During the 10 days treatment period and the 3 months follow-up period.
  The antibacterial application time of each group of subjects was counted.
Endotracheal intubation rate | In 10 days of the treatment period.
  The number of endotracheal intubation cases in the two groups during the treatment period was calculated.
Case fatality rate | During the 10 days treatment period and the 3 months follow-up period.
  The number of deaths due to AECOPD in the two groups during the study period was counted.

IPD SHARING:
Plan to Share IPD: No